CLINICAL TRIAL: NCT06062199
Title: Impact of Implementing the Modified A-DIVA Scale on Successful Access to a Venous Line on the First Attempt
Acronym: DIVAPERF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 2023-A01480-45
Record Dates: First submitted 2023-09-25; First posted 2023-10-02 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control arm (No Intervention): Nurses will place a peripheral venous line on these patients without having been trained in the venous status score predictive of failure.
- Experimental arm (Experimental): Nurses will place a peripheral venous line on these patients after being trained in the venous status score predictive of failure.
  Interventions: Procedure: Training in the A-DIVA scale and its failure prediction score

INTERVENTIONS:
Procedure: Training in the A-DIVA scale and its failure prediction score — Nurses are trained in the A-DIVA scale and its predictive failure score. This score enables them to adapt their approach to peripheral venous line insertion.
  Arms: Experimental arm

SUMMARY:
Peripheral venous access (PVA), although commonly used, can be a difficult procedure for patients with precarious venous capital. The difficulty of insertion can lead to multiple attempts, with the consequences of pain, anxiety, delayed management and worsening of the potentially already precarious venous capital. One study assessed the risk of failure according to a score based on venous status criteria. This study first established a link between venous status criteria and the risk of failure. The criteria defined as determinants were used to establish a venous status score. The data were then repeated by analyzing the success rate as a function of the scale score. A clear link between score and risk of failure was established. It seems worthwhile to evaluate the impact of implementing this scale prior to the placement of a peripheral venous line.

The hypothesis is that obtaining a score predictive of failure would modify the therapeutic attitude of the registered nurse. They would opt for techniques that would increase their chances of success. This in turn would lead to a reduction in unsuccessful attempts, which generate pain and anxiety for the patient. Preserving venous capital by increasing first-attempt success is both a health issue for the patient and a guarantee of quality of care.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient of legal age included in a care program requiring a VVP;
* Fluency in French
* Patient affiliated to a social security scheme;
* Written, signed and dated informed consent.

Exclusion Criteria:

* As the A-DIVA scale specifies a search for venous access to the upper limb, any patient without an upper limb or with a condition that contraindicates VVP placement in the upper limbs will be excluded;
* Patients treated as emergencies;
* Patients with a language barrier or known significant cognitive or psychiatric disorders;
* Patients under guardianship, curatorship, deprivation of liberty or legal protection;
* Pregnant or breast-feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Success rate of peripheral venous vein placement | 1 year
  Success rate of peripheral venous vein insertion on the first attempt in the 2 groups (group in which VVP insertion will be performed by nurses not trained in the A-DIVA score and group in which VVP insertion will be performed after score assessment by nurses trained in the A-DIVA score) expressed by the number of attempts equal to 1.

SECONDARY OUTCOMES:
Total number of attempts | 1 year
  Total number of attempts
Number of visualization techniques, alternative devices and/or third-party assistance used | 1 year
  Number of visualization techniques, alternative devices and/or third-party assistance used
Pain score: Numerical Pain Scale | 1 year
  The pain score is based on a numerical pain scale ranging from 0 to 10, with 0 representing no pain and 10 representing unbearable pain.
Number of years' experience of nurses since obtaining diploma in nursing | 1 year
  Number of years' experience of nurses since obtaining diploma in nursing
A-DIVA scale score | 1 year
  The A-DIVA score (Adult Difficult Intravenous Access Score) predicts the difficulty of infusing an adult. The score ranges from 0 to 5, with 0 being the lowest risk of difficulty, and 5 being the highest.

CONTACTS AND LOCATIONS:
Overall Officials: Lucie MADELAINE, Study Director — Centre Jean Perrin
Locations (3):
- France (3):
  - CHU Gabriel Montpied, Clermont-Ferrand
  - Centre Jean PERRIN, Clermont-Ferrand
  - Hôpital de la Croix Rousse, Lyon

IPD SHARING:
Plan to Share IPD: Undecided